CLINICAL TRIAL: NCT04911322
Title: Correlation Between Pulmonary Artery Doppler And Other Ultrasonographic Markers With Neonatal Outcome In Placenta Accreta Spectrum Patients
Brief Title: Pulmonary Artery Doppler and Neonatal Outcome in Placenta Accreta Spectrum Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noran Amin, Nominated demonstrator of Obstetrics and Gynecology, Cairo University, Cairo University
Other Study IDs: PAS disorders
Record Dates: First submitted 2021-05-23; First posted 2021-06-03 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasonography — A full obstetric ultrasound scan will be performed to assess signs of placental invasion, to document fetal biometry, estimated fetal weight, amniotic fluid index, assess fetal lung maturity parameters as pulmonary artery Doppler waveforms, amniotic fluid free floating particles, bowel echogenicity, fetal epiphyseal ossific centers, liver/lung echogenicity and kidney length.
  Pulmonary artery Doppler: Fetal echocardiography will be done. Pulmonary artery Doppler ﬂow waveforms, including pulsatility index, resistance index, systolic-to-diastolic ratio, peak systolic velocity, and acceleration time to ejection time ratio will be measured in the main pulmonary artery.

SUMMARY:
To correlate ultrasonographic markers of fetal lung maturity including Pulmonary artery Doppler indices in the late preterm and early term in placenta accreta spectrum patients with neonatal outcome.

DETAILED DESCRIPTION:
The increasing rates of cesarean section has led to several fold increase in the incidence of placenta accreta spectrum in the last three or four decades.

Placenta accreta spectrum (PAS) disorders is the term used to describe a variety of pregnancy complications resulting from abnormal placental implantation that is accompanied by deﬁciency of the uterine wall.

Placenta accreta spectrum includes placenta accreta, placenta increta, placenta percreta.

Placenta accreta spectrum is one of the devastating obstetric complications owing to massive hemorrhage encountered during manual removal of the placenta to preserve the uterus or even the need for peripartum hysterectomy, need for massive blood transfusion, maternal intensive care admission and maternal mortality.

Complications related to blood loss are lower in elective compared to emergency deliveries. This has led to the scheduling of surgical interventions with planned late preterm (35-36 weeks) or early term (37 weeks) delivery as a mechanism to avoid the need for emergency surgery. According to the RCOG guidelines, planned delivery at 35 0/7- 36 0/7 weeks of gestation provides the best chance between fetal maturity and the risk of unscheduled delivery while ACOG recommends 34 0/7- 35 6/7.

Early attempts have been made to predict fetal maturity on the basis antenatal sonographic parameters including lung characteristics, bowel pattern, placental grading (which cannot be relied upon in patients with placenta accreta spectrum), and the presence or absence of intraamniotic particles (vernix caseosa).

Additionally, the epiphyseal ossification centers appear and enlarge at variable rates but in a predictable sequence: the distal femoral epiphysis (DFE) appears prior to the proximal tibial epiphysis (PTE), which precedes the appearance of the proximal humeral epiphysis (PHE). The PTE grows more rapidly than does the DFE so that, as gestation progresses, the size of the PTE approaches that of the DFE.

More recently, fetal pulmonary artery Doppler has been used to predict neonatal RDS. It was found that an elevated acceleration-to-ejection time ratio was significantly associated with neonatal RDS. However such indices cannot be generalized in all cases, especially those with placenta accreta spectrum who have excessive placental shunting affecting fetoplacental circulation resistance.

To the best of our knowledge, no available studies have correlated signs of maturity of the fetus detected by ultrasound with neonatal outcomes in the late preterm and early term in such patients. Presence of such signs of maturity can aid the obstetrician to choose the most appropriate timing for termination especially in low income countries who have limited access to NICUs.

Being cost effective and non invasive, ultrasonography is used as a routine obstetric scanning tool. This study will help determine the utility of ultrasound in assessing the fetal lung maturity in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-42 years old
* Patients who will be diagnosed with placenta accreta spectrum preoperatively according to (ACOG 2018), (Jauniaux et al., 2018 a), (Jauniaux et al., 2018 b)
* Those who will undergo elective or emergency cesarean.
* With gestational age: 34 0/7 - 38 6/7 weeks
* Under the effect of general anesthesia

Exclusion Criteria:

* Multifetal pregnancy
* Intrauterine fetal death
* Intrauterine growth restriction (IUGR) which is defined as a rate of fetal growth that is less than normal for the growth potential of that specific infant
* Diabetes with pregnancy either gestational or overt which is defined as any degree of glucose intolerance with an onset or first recognition during pregnancy
* Pregnancy induced hypertension defined as either systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg. It is classified as one of four conditions: preexisting hypertension, gestational hypertension, preeclampsia, preexisting hypertension with superimposed preeclampsia
* Premature rupture of membranes
* BMI above 40 due to technical difficulties to obtain accurate measures
* Narcotic usage during anesthesia before fetal delivery
* Major congenital fetal anomalies whether diagnosed before or after delivery
* Maternal fever more than 37.4 degree
* Emergent cases presenting with fetal distress (bradycardia will be defined as fetal heart rate < 110 beat per minute)
* Patients who have not completed the course of antenatal corticosteroids according to (RCOG 2010).
* Intraoperative spontaneous separation of the placenta

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Women with placenta accreta spectrum with singleton pregnancy undergoing cesarean delivery in Kasr Alainy hospital.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Acceleration time to ejection time (At/Et) ratio of fetal pulmonary artery Doppler in neonates with good and poor outcome. | Baseline
  (At/Et) ratio will be measured in the fetal main pulmonary artery Doppler and will be correlated with the neonatal outcome

SECONDARY OUTCOMES:
The pulsatility index (PI) of the fetal pulmonary artery Doppler in neonates with good and poor outcome. | Baseline
  The PI will be measured in the fetal main pulmonary artery and will be correlated with the neonatal outcome
The resistance index (RI) of the fetal pulmonary artery Doppler in neonates with good and poor outcome | Baseline
  RI will be measured in the fetal main pulmonary artery and will be correlated with the neonatal outcome
The systolic to diastolic ratio (S/D) of the fetal pulmonary artery Doppler in neonates with good and poor outcome | Baseline
  S/D will be measured in the fetal main pulmonary artery and will be correlated with the neonatal outcome
The peak systolic velocity (PSV) of the fetal pulmonary artery Doppler in neonates with good and poor outcome | Baseline
  PSV will be measured in the fetal main pulmonary artery and will be correlated with the neonatal outcome
Optimal timing of delivery in PAS for best neonatal outcome | baseline
  according to the neonatal outcome, the best timing for delivery will be determined
Optimal timing of delivery in PAS for best maternal outcome | baseline
  according to the maternal mortality and morbidity rate, the best timing for delivery will be obtained
percent of women who will undergo cesarean hysterectomy versus conservative management | baseline
  surgical management options; cesarean hysterectomy and conservative management will be recorded
The need for blood transfusion | baseline
  The need for replacement by blood or blood products will be recorded
Maternal morbidity in the form of organ injury will be recorded | baseline
  Organ injury will be recorded
The need for peripartum hysterectomy will be recorded | Baseline
  The need for peripartum hysterectomy either in cases of abnormally invasive placenta or in cases of abnormally adherent placenta in which the placenta separated but with uncontrollable bleeding
Maternal mortality rate | Baseline
  Rate of maternal mortality will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H El Sawaf, MD, Study Director — Cairo University; Tarek M El Husseiny, MD, Study Chair — Cairo University
Locations (1):
- Kasralainy Cairo University, Giza, Egypt

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists; Society for Maternal-Fetal Medicine. Obstetric Care Consensus No. 7: Placenta Accreta Spectrum. Obstet Gynecol. 2018 Dec;132(6):e259-e275. doi: 10.1097/AOG.0000000000002983. PMID 30461695
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Buchanan TA, Xiang AH. Gestational diabetes mellitus. J Clin Invest. 2005 Mar;115(3):485-91. doi: 10.1172/JCI24531. PMID 15765129
- [Background] Hobson SR, Kingdom JC, Murji A, Windrim RC, Carvalho JCA, Singh SS, Ziegler C, Birch C, Frecker E, Lim K, Cargill Y, Allen LM. No. 383-Screening, Diagnosis, and Management of Placenta Accreta Spectrum Disorders. J Obstet Gynaecol Can. 2019 Jul;41(7):1035-1049. doi: 10.1016/j.jogc.2018.12.004. PMID 31227057
- [Background] Creanga AA, Bateman BT, Butwick AJ, Raleigh L, Maeda A, Kuklina E, Callaghan WM. Morbidity associated with cesarean delivery in the United States: is placenta accreta an increasingly important contributor? Am J Obstet Gynecol. 2015 Sep;213(3):384.e1-11. doi: 10.1016/j.ajog.2015.05.002. Epub 2015 May 5. PMID 25957019
- [Background] Eller AG, Porter TF, Soisson P, Silver RM. Optimal management strategies for placenta accreta. BJOG. 2009 Apr;116(5):648-54. doi: 10.1111/j.1471-0528.2008.02037.x. Epub 2009 Feb 4. PMID 19191778
- [Background] Hornberger LK, Sahn DJ. Rhythm abnormalities of the fetus. Heart. 2007 Oct;93(10):1294-300. doi: 10.1136/hrt.2005.069369. No abstract available. PMID 17890709
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097
- [Background] Jauniaux E, Bhide A, Kennedy A, Woodward P, Hubinont C, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Prenatal diagnosis and screening. Int J Gynaecol Obstet. 2018 Mar;140(3):274-280. doi: 10.1002/ijgo.12408. No abstract available. PMID 29405319
- [Background] Kim SM, Park JS, Norwitz ER, Hwang EJ, Kang HS, Park CW, Jun JK. Acceleration time-to-ejection time ratio in fetal pulmonary artery predicts the development of neonatal respiratory distress syndrome: a prospective cohort study. Am J Perinatol. 2013 Nov;30(10):805-12. doi: 10.1055/s-0032-1333132. Epub 2013 Jan 4. PMID 23292917
- [Background] Mahony BS, Bowie JD, Killam AP, Kay HH, Cooper C. Epiphyseal ossification centers in the assessment of fetal maturity: sonographic correlation with the amniocentesis lung profile. Radiology. 1986 May;159(2):521-4. doi: 10.1148/radiology.159.2.3515425.
- [Background] Mammaro A, Carrara S, Cavaliere A, Ermito S, Dinatale A, Pappalardo EM, Militello M, Pedata R. Hypertensive disorders of pregnancy. J Prenat Med. 2009 Jan;3(1):1-5. PMID 22439030
- [Background] McCowan LM, Figueras F, Anderson NH. Evidence-based national guidelines for the management of suspected fetal growth restriction: comparison, consensus, and controversy. Am J Obstet Gynecol. 2018 Feb;218(2S):S855-S868. doi: 10.1016/j.ajog.2017.12.004. PMID 29422214
- [Background] Seoud MA, Nasr R, Berjawi GA, Zaatari GS, Seoud TM, Shatila AS, Mirza FG. Placenta accreta: Elective versus emergent delivery as a major predictor of blood loss. J Neonatal Perinatal Med. 2017;10(1):9-15. doi: 10.3233/NPM-1622. PMID 28304318
- [Background] Spong CY, Mercer BM, D'Alton M, Kilpatrick S, Blackwell S, Saade G. Timing of indicated late-preterm and early-term birth. Obstet Gynecol. 2011 Aug;118(2 Pt 1):323-333. doi: 10.1097/AOG.0b013e3182255999. PMID 21775849
- [Background] Varner S, Sherman C, Lewis D, Owens S, Bodie F, McCathran CE, Holliday N. Amniocentesis for fetal lung maturity: will it become obsolete? Rev Obstet Gynecol. 2013;6(3-4):126-34. PMID 24826202
- [Background] Warshak CR, Ramos GA, Eskander R, Benirschke K, Saenz CC, Kelly TF, Moore TR, Resnik R. Effect of predelivery diagnosis in 99 consecutive cases of placenta accreta. Obstet Gynecol. 2010 Jan;115(1):65-69. doi: 10.1097/AOG.0b013e3181c4f12a. PMID 20027036
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Gyamfi-Bannerman C. Society for Maternal-Fetal Medicine (SMFM) Consult Series #44: Management of bleeding in the late preterm period. Am J Obstet Gynecol. 2018 Jan;218(1):B2-B8. doi: 10.1016/j.ajog.2017.10.019. Epub 2017 Oct 25. PMID 29079144